CLINICAL TRIAL: NCT03798756
Title: Automated Check-in Data Collection Study
Acronym: ACDC
Status: Completed | Type: Observational
Sponsor: Keele University (Other)
Responsible Party: Sponsor
Other Study IDs: RG-0275-18 V1.0
Record Dates: First submitted 2018-09-14; First posted 2019-01-10 (Actual); Results first posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-03

CONDITIONS: Primary Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to examine patient acceptability, for providing brief research information, whilst self-completing an automated check-in screen prior to any general practice consultation.

DETAILED DESCRIPTION:
The Automated Check-in Data Collection (AC DC) Study, is a pilot feasibility study, observing patients consulting in general practice and completing an automated check-in screen prior to their booked appointment, to confirm their attendance. Participants will be recruited over three weeks from approximately 11 participating general practices.

The primary objective of the study is to assess patient acceptability for answering brief research questions in the general practice waiting room, using an automated check-in screen. This will be measured by observing the percentage of completed automated check-in screens with entered research data.

Secondary objectives will assess check-in completion of self-reported pain and willingness to be contacted about future research studies of relevance. Reported severity of bodily pain experienced over the last 4 weeks and the proportion of patients agreeing to be contacted about future research studies of relevance, will be observed.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or over attending participating general practices for a consultation with any healthcare professional.
* Patients registered with the participating general practice during the specified recruitment period.
* Patients able to read and respond in English.

Exclusion Criteria:

• Patients under the age of 18 attending the general practice for a consultation with a healthcare professional.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients of age 18 and over, who can read and respond in English and with a booked appointment, consulting with any Health Care Professional (HCP) at their general practice, during the recruitment period will be eligible to participate. All patients are required to confirm their attendance at the general practice by using the automated check-in screen. If the patient completing the automated check-in screen is 18 years of age or over, the additional two research questions will appear for completion.
Sampling Method: Probability Sample
Enrollment: 9274 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-04-14 (Actual); Study Completion 2019-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian D Mallen, Study Director — University of Keele
Locations (1):
- New Cross Hospital, Wolverhampton, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort: Automated check-in
Period: Overall Study
Arm/Group | Cohort
Started | 9274
Completed | 9274
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort: This was a Cohort, there were no arms. It was an entire group.
Arm/Group | Cohort
Number analyzed (Participants) | 9274
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5982
  >=65 years | 3292
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5653
  Male | 3621
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 9274
Patients checking in for a consultation, answering a research question, using check-in sceen [Count of Participants; unit: Participants] | 9274

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Bodily Pain
Description: To assess what self-reported degrees of pain were reported by participants and what proportion of participants did answer a research question within the general practice waiting room using an automated check-in screen.
Time Frame: Through study completion at 1st visit (Day 1)
Measure: Count of Participants; unit: Participants
Groups:
- Bodily Pain: To assess patient acceptability of answering a research question on bodily pain, in the general practice waiting room using an automated check-in screen.
Arm/Group | Bodily Pain
Number analyzed (Participants) | 9274
Participants
  None | 2937
  Very mild | 1061
  Mild | 1446
  Moderate | 2344
  Severe | 1125
  Very Severe | 9
  Not documented | 352

2. Secondary Outcome: Bodily Pain Response
Description: Proportion of participants answering the bodily pain research question using an automated check-in screen.
Time Frame: Through study completion at 1st visit (Day 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort
Number analyzed (Participants) | 9274
Participants | 8922

3. Secondary Outcome: Consent to Contact Response
Description: Proportion of participants answering the consent to contact research question using an automated check-in screen.
Time Frame: Through study completion at 1st visit (Day 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Bodily Pain
Number analyzed (Participants) | 9274
Participants | 8285

ADVERSE EVENTS:
Groups:
- Cohort: All those patients checking-in for a pre-booked consultation using an automated check-in screen and answering at least one research question
Arm/Group | Cohort
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/56/NCT03798756/Prot_SAP_000.pdf